CLINICAL TRIAL: NCT01692392
Title: Short and Long-term Effects of Surgical Repair of Pectus Carinatum - A Questionnaire Study of Health-related Quality of Life, Persisten Post-surgical Pain and Sensory Disturbances.
Brief Title: Health-related Quality of Life in Patients Undergoing Surgery for Pectus Carinatum
Acronym: HRQoL
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PECCAR-1
Record Dates: First submitted 2012-09-12; First posted 2012-09-25 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2012-09

CONDITIONS: Pectus Carinatum; Quality of Life; Pain, Postoperative; Somatosensory Disorders
Keywords: Pectus carinatum; Quality of life; Pain, postoperative; Somatosensory disorders
MeSH Terms: conditions — Pectus Carinatum; Pain, Postoperative; Somatosensory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pectus carinatum: Patients who have undergone surgical repair of pectus carinatum.

SUMMARY:
The purpose of the study is to assess changes in health-related quality of life in patients undergoing surgical correction of pectus carinatum. In addition, the study assessed long-term effects of surgical intervention in relation to the development of persistent postoperative pain and / or sensory disturbances in the surgical field.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgery for pectus carinatum

Exclusion Criteria:

* patients without pectus carinatum

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients referred to the Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby for the purpose of surgery for pectus carinatum from May 1, 2012 to May 1, 2013 are invited to participated in the study
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in health-related quality of life at 6 months | From baseline (the day before surgery) to six month follow-up (six months after surgery)
  Health-related Quality of Life (HRQoL) will be assessed by means of a validated Danish version of the Short-Form 36 Health Survey (SF-36)

SECONDARY OUTCOMES:
Persistent post-surgical pain | Six month following surgery
  In this study persistent post-surgical pain is defined as pain developing after pectus surgery and lasting for at least 4 months. Other causes of pain (e.g. infection) and pain continuing from a pre-existing pain problem will be excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Skejby, Department of Cardiothoracic and Vacular Surgery, Aarhus, Denmark